CLINICAL TRIAL: NCT06067815
Title: Assessment of Right Ventricular Function in Patient With Severe Mitral Stenosis Before and After Balloon Mitral Valvuloplasty
Brief Title: Assessment of Right Ventricular Function in Patients With Severe Mitral Stenosis Before and After Balloon Mitral Valvuloplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yassmin Zakaria Basheir, Assessment of right ventricular function in patient with severe mitral stenosis before and after balloon mitral valvuloplasty, Assiut University
Other Study IDs: Mitral stenosis PTMC
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Mitral Stenosis
MeSH Terms: conditions — Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To detect short-term impacts of successful balloon mitral valvuloplasty on right ventricular function

DETAILED DESCRIPTION:
In patients with mitral valve stenosis, right ventricular failure may develop either by the rheumatic process directly or through hemodynamic alterations resulting from pulmonary vascular changes.

Right ventricular (RV) function plays an important role in development of clinical symptoms and prognosis in patients with mitral stenosis (MS).This is primarily affected by hemodynamic effects on RV due to pulmonary hypertension(PH).

In the last two decades, Percutaneous Transluminal Mitral Commissurotomy (PTMC) has become the treatment of choice for patients with symptomatic rheumatic MS . Using this method,Mitral Valve Area (MVA) can be increased, which can improve the hemodynamic and clinical features of patients with MS .

RV functional assessment is difficult and not done routinely because of its complex anatomy and high load dependence.

Different modalitis are used to assess RV function as Tissue Doppler and two-dimensional (2D) speckle tracking method has been used to quantify strain for assessment Myocardial strain is a measure of tissue deformation, which is expressed as a percentage change.

ELIGIBILITY:
Inclusion Criteria:

* Patient with isolated mitral stenosis (except those with mild mitral regurgitation and are candidate for PTMC by 2D Echo evaluation).

  * Patient with normal left ventricular EF.
  * patient with sinus rhythm or AF
  * patient with any degree of pulmonary HTN

Exclusion Criteria:

* Patient with another valve lesion or more than mild mitral regurgitation.
* Patient with impaired cardiac function.
* patient with coronary arteries disease
* Mitral stenosis of other etiology than rheumatic origin.

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe mitral stenosis,not impairment left ventricular function
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
To compare RV function before and after PTMC | 1 year
  echocardiogram

SECONDARY OUTCOMES:
To measure the right side pressure changes invasively before and after PTMC | 1 year
  Right sided heart catheterization
To compare the effect of PTMC on RV function in patient with AF and sinus rythm | 1year

REFERENCES:
- [Background] Kumar V, Jose VJ, Pati PK, Jose J. Assessment of right ventricular strain and strain rate in patients with severe mitral stenosis before and after balloon mitral valvuloplasty. Indian Heart J. 2014 Mar-Apr;66(2):176-82. doi: 10.1016/j.ihj.2014.02.012. Epub 2014 Mar 1. PMID 24814111